CLINICAL TRIAL: NCT04183660
Title: A Post Market Surveillance Study of the Hemovent Extracorporeal Cardiopulmonary Support System for Cardiac and Respiratory Support: The MOBYBOX Trial
Brief Title: A Post Market Surveillance Study of the Hemovent Extracorporeal Cardiopulmonary Support System:The MOBYBOX Trial
Status: Recruiting | Type: Observational
Sponsor: Hemovent GmbH (Industry)
Collaborators: seleon GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: HVT-MB1
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Failure; Respiratory Failure; Cardio-Respiratory Failure; Imminent Cardiorespiratory or Respiratory Failure
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MOBYBOX System — extracorporeal cardiopulmonary support

SUMMARY:
The purpose of this study is to evaluate prospectively the safety and performance of the MOBYBOX System in the veno-arterial configuration in patients with cardiorespiratory failure or in the veno-venous configuration in patients with severe respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cardiac, respiratory or cardiorespiratory failure or imminent failure and 1 of the 5 following sets of findings:

  1. A Murray score ≥ 3.0 and/or severe hypoxemia with A PaO2/FIO2 > 100 mm on 0.9 FIO2;
  2. Uncompensated hypercapnia with pH <7.2 despite a Pplateau > 30 cm H20;
  3. Significant air leak/bronchopleural fistula;
  4. Need for intubation in a patient on lung transplant list;
  5. Immediate/risk of cardiac or respiratory collapse (pulmonary embolus, blocked airway, blocked blood flow, unresponsive to optimal care);
* Written consent of the patient or the legal guardian or external consulting physician as designated and approved by the Ethics Committee.

Exclusion Criteria:

* High pressure ventilation (FIO2 > 0.9 and Pplateau > 30 cm H2O) or high FIO2 requirements for more than 7 days;
* Severe intracranial bleeding, which precludes the use of anticoagulation therapy or any other inability to be anticoagulated
* Excessive weight (> 180 Kg)
* Severe irreversible brain injury (e.g., hypoxic brain injury)
* Inability to accept blood products;
* Any condition or organ dysfunction that would limit the likelihood of overall benefit from ECMO, such as severe, irreversible brain injury, hepatic and/or renal failure, or untreatable metastatic cancer;
* Immunosuppression with an absolute neutrophil count < 400/mm3;
* Patient has been treated with ECMO ≤ 48 hours.
* For veno-veno ECMO in the setting of respiratory failure the following exclusion criteria apply:
* Severe pulmonary hypertension (mPAP > 50 mm Hg)
* Severe right or left sided heart failure (EF < 25%)
* For veno-arterial ECMO in the setting of cardiac insufficiency:
* Severe aortic regurgitation
* Aortic dissection.
* The patient is moribund, or the patient has severe or deteriorating damage in critical body systems.
* Patient is participating in an investigational drug or device study trial that has not reached the primary endpoint or that interferes with the current study endpoints.
* Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consented patients with cardiorespiratory failure or ith severe respiratory failure who meet all of the inclusion and none of the exclusion criteria and in whom the investigator intends to treat the patient with cardiopulmonary support using the Hemovent MOBYBOX System.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rates of device and procedure related serious adverse events | 24 hours
  Acute safety defined as rates of device and procedure related serious adverse events up to 24 hours post-intervention.

SECONDARY OUTCOMES:
Device performance success | every 4 hours while the patient receives ECMO using the MOBYBOX device
  Device performance success (defined as the ability to establish either veno-arterial ECMO to support cardiorespiratory function and tissue oxygenation or veno-venous ECMO to support respiratory function and tissue oxygenation)
Adverse Event rate | 24 hours
  Acute safety defined as rates adverse events up to 24 hours post-intervention.
Mortality rate | 30 days
  All-cause mortality up to 30 days post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, Prof., Principal Investigator — Uniklinikum Essen
Locations (4):
- Germany (4):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Helios Klinikum Erfurt, Erfurt